CLINICAL TRIAL: NCT00368914
Title: Pharmacodynamic-Guided Dose Finding Study of Rapamycin (Rapamune®, Sirolimus) in Adult Patients With Solid Tumors
Brief Title: Sirolimus in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: JHOC-J0402, CDR0000491204; R21CA112919 (NIH); P30CA006973 (NIH); JHOC-J0402; JHOC-04032602
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Sirolimus; Biopsy

INTERVENTIONS:
Drug: sirolimus
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of sirolimus in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacodynamic optimal dose of sirolimus, by evaluating p70^s6 kinase inhibition in peripheral blood mononuclear cells (PBMC) and normal skin, in patients with metastatic or unresectable solid tumors.
* Correlate target inhibition in tumor tissue with PBMC and normal skin target inhibition in patients whose tumors are amenable to sequential tumor biopsies.

Secondary

* Characterize the pharmacokinetics of sirolimus in these patients
* Determine the pharmacodynamic effects of sirolimus on tumor, normal skin, and normal oral mucosa of these patients
* Correlate the pharmacodynamic effects of sirolimus with pharmacokinetics and clinical effects.
* Correlate the Akt signaling pathway with pharmacodynamic endpoints.
* Explore pharmacokinetic-pharmacodynamic and toxicodynamic relationships of sirolimus in these patients.
* Quantify the toxicity of sirolimus in these patients.
* Evaluate, preliminarily, the activity of sirolimus in these patients.

OUTLINE: This is a prospective, dose-escalation study.

Patients receive oral sirolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. The pharmacodynamic optimal dose is considered the dose at which 10 patients are treated without requiring further dose escalation.

Patients undergo blood collection, tumor tissue and normal skin biopsies, and oral mucosal smears periodically for pharmacodynamic, pharmacokinetic, and biomarker correlative studies.

After completion of study treatment, patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor malignancy

  * Metastatic or inoperable disease
  * Failed curative or standard palliative therapy OR no such therapy exists
* Evaluable or measurable disease

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Tumor amenable to serial biopsies
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG 0-1
* Life expectancy ≥ 3 months
* WBC > 3,500/mm³
* Absolute neutrophil count > 1,500/mm³
* Hemoglobin > 9 g/dL
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2 mg/dL
* ALT and AST ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Triglycerides < 2 times ULN
* Total cholesterol < 2 times ULN
* Willing to undergo serial tumor biopsies and normal skin biopsies
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No immunodeficiency
* No gastrointestinal tract disease resulting in an inability to take oral medication
* No requirement for IV alimentation
* No active peptic ulcer disease
* No active infections
* No other uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this therapy
* No concurrent or second malignancy within the past 5 years
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 12 months
  * Unstable angina
  * Peripheral vascular disease ≥ grade 2
  * Uncontrolled congestive heart failure
  * Uncontrolled hypertension (i.e., systolic blood pressure [BP] > 170 mm Hg, diastolic BP > 95 mm Hg)

PRIOR CONCURRENT THERAPY:

* Recovered from prior anticancer therapy

  * No unresolved chronic toxicity > CTC grade 2
* No prior surgical procedures affecting absorption
* More than 4 weeks since prior surgery except minor procedures (e.g., dental work or skin biopsy)
* More than 1 month since prior participation in an investigational drug trial
* More than 1 month since prior chemotherapy
* No concurrent use of any of the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Cyclosporine
  * Clarithromycin
  * Diltiazen
  * Clotrimazole
  * Ketoconazole
  * Fluconazole
  * Hypericum perforatum (St. John's wort)
  * Cimetidine
  * Grapefruit juice
* No concurrent immunosuppressants
* No other concurrent investigational or commercial agents or therapies for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic optimal dose of sirolimus by evaluation of p70s6 kinase inhibition in peripheral blood mononuclear cells (PBMC) and normal skin
Correlation of target tissue inhibition in tumor tissue with PMBCs and normal skin

SECONDARY OUTCOMES:
Pharmacokinetics
Pharmacodynamic effects of sirolimus on tumor, normal skin, and normal oral mucosa
Correlation of pharmacodynamic effects of sirolimus with pharmacokinetics and clinical effects
Pharmacokinetic-pharmacodynamic and toxicodynamic relationships
Correlation of activation of the mTOR pathway in tumor tissue with the antitumor effects of sirolimus
Toxicity by NCI Common Toxicity Criteria Version 3.0
Activity of sirolimus
Response rate by RECIST criteria
Overall survival and progression-free survival by Kaplan-Meier method at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Jimeno A, Rudek MA, Kulesza P, Ma WW, Wheelhouse J, Howard A, Khan Y, Zhao M, Jacene H, Messersmith WA, Laheru D, Donehower RC, Garrett-Mayer E, Baker SD, Hidalgo M. Pharmacodynamic-guided modified continuous reassessment method-based, dose-finding study of rapamycin in adult patients with solid tumors. J Clin Oncol. 2008 Sep 1;26(25):4172-9. doi: 10.1200/JCO.2008.16.2347. PMID 18757332